CLINICAL TRIAL: NCT02747407
Title: Determining the Competence of the Immune System Over the First Year of Therapy in Patients With Glioma: A Battery of Quantitative, Qualitative and Functional Measures of Immune Readiness
Brief Title: Qualitative, Qualitative, and Functional Studies Over the First Year in Measuring Immune System Response During the First Year of Therapy in Patients With Brain Tumors
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00037250; NCI-2016-00472 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU 01316 (Other: Comprehensive Cancer Center of Wake Forest University); P30CA012197 (NIH)
Record Dates: First submitted 2016-04-19; First posted 2016-04-21 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Astrocytoma; Glioma; Oligodendroglioma
MeSH Terms: conditions — Astrocytoma; Glioma; Oligodendroglioma | interventions — Hepatitis A Vaccines; Tetanus Toxoid; Influenza Vaccines; fluarix; FluBlok; FluLaval

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — peripheral blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Basic Science Group II (vaccination at 9 months): Patients undergo standard of care treatment and collection of blood samples as in Group I. Patients then receive hepatitis A and tetanus toxoid vaccinations at month 9.
  Interventions: Biological: Hepatitis A Vaccine; Other: Laboratory Biomarker Analysis; Biological: Tetanus Toxoid Vaccine; Biological: Trivalent Influenza Vaccine
- Basic Science Groups I (vaccination pre-treatment): Patients receive standard of care hepatitis A or B vaccine, tetanus toxoid vaccine, and trivalent influenza vaccine and then undergo standard of care treatment external beam radiation therapy and receive standard of care temozolomide. Patients also undergo collection of blood Samples monthly for the first 8 months and then bimonthly for up to 12 months for analysis via flow cytometry, (CFSE) assay, live cell/dead cell distinction assay, and determination of naïve and memory immune response.
  Interventions: Biological: Hepatitis A Vaccine; Other: Laboratory Biomarker Analysis; Biological: Tetanus Toxoid Vaccine; Biological: Trivalent Influenza Vaccine

INTERVENTIONS:
Biological: Hepatitis A Vaccine
  Other Names: Havrix; Hepatitis A Vaccine, Inactivated; Vaqta
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Tetanus Toxoid Vaccine
  Other Names: Tetanus Toxoid; TT
Biological: Trivalent Influenza Vaccine
  Other Names: Agriflu; Flu prevention; Flu prophylaxis; Flu shot; Flu vaccination; Fluarix; Flublok; FluLaval; Flushield; Fluvirin; Fluzone; Influenza Vaccine; Influenza Virus Vaccine, Trivalent, Types A and B; TIV

SUMMARY:
This research trial studies qualitative, qualitative, and functional studies over the first year in measuring immune system response in patients with brain tumors. Measuring the number of immune cells, whether these immune cells work correctly, and response to 2 vaccines at several times during the first year of treatment may help find out how active the immune system responds to fight infection and cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To describe the quantity of immune cells underlying the antitumor immune response including dendritic cells, naive and activated T- and B-cells, regulatory T-cells, and natural killer cells.

II. To determine the proliferative ability of lymphocytes via T-cell activation.

SECONDARY OBJECTIVES:

I. To describe the immunologic response to the hepatitis A vaccine (or hepatitis B vaccine in those who are hepatitis A exposed) in comparison to expected/known normal responses either prior to (i.e. pre-treatment) or following chemoradiation (i.e. post-treatment).

II. To describe the immunologic response to tetanus toxoid vaccination compared to expected/known normal responses either prior to (i.e. pre-treatment) or following chemoradiation (i.e. post-treatment).

TERTIARY OBJECTIVES:

I. To describe the immunologic response to the yearly influenza vaccination over the course of the first year of therapy for glioma (timing of administration will be when clinically indicated over this year of therapy).

II. To describe the frequency of viral infection in glioma patients hospitalized during the respiratory viral season within year 1 of therapy.

III. To describe the overall survival of glioma patients enrolled in this study and describe the overall survival in these patients by changes in immunologic function.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I: Patients receive standard of care hepatitis A or B vaccine, tetanus toxoid vaccine, and trivalent influenza vaccine and then undergo standard of care treatment external beam radiation therapy and receive standard of care temozolomide. Patients also undergo collection of blood Samples monthly for the first 8 months and then bimonthly for up to 12 months for analysis via flow cytometry, carboxyfluorescein diacetate succinimidyl ester (CFSE) assay, live cell/dead cell distinction assay, and determination of naïve and memory immune response.

GROUP II: Patients undergo standard of care treatment and collection of blood samples as in Group I. Patients then receive hepatitis A and tetanus toxoid vaccinations at month 9.

ELIGIBILITY:
Inclusion Criteria:

* Clinically or histologically diagnosed primary central nervous system astrocytoma or oligodendroglioma of World Health Organization grade II, III or IV
* Anticipated to undergo treatment with concurrent chemoradiation with conformal external beam radiotherapy in combination with low-dose temozolomide (75 mg/m^2) followed by adjuvant temozolomide (150-200 mg/m^2)
* Able to provide informed consent
* Karnofsky performance status >= 50%
* Willing and able to receive the tetanus toxoid and hepatitis vaccination (though prior vaccination with either vaccine is not a contraindication to eligibility)

Exclusion Criteria:

* Concurrent enrollment on an experimental study involving an agent whose primary mechanism of action is the immune system (i.e. immune checkpoint inhibition, oncologic vaccine, or other immune-directed therapies); Note: patients enrolled on an experimental study or receiving another concurrent treatment in addition to standard chemoradiation whose primary mechanism of action is NOT the immune system will be eligible for enrollment
* Patients unable to receive tetanus toxoid vaccination

  * Guillain-Barré syndrome =< 6 weeks after previous dose of a tetanus toxoid-containing vaccine; unstable neurologic condition (e.g., cerebrovascular events and acute encephalopathic conditions) which does not include the patient's primary brain tumor; history of an Arthus reaction following a previous dose of a tetanus toxoid-containing and/or diphtheria toxoid-containing vaccine
* Patients unable to receive hepatitis vaccination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with primary central nervous system astrocytoma or oligodendroglioma
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2021-09-09 (Actual)

PRIMARY OUTCOMES:
Proliferative ability of lymphocytes by carboxyfluorescein diacetate succinimidyl ester assay | Up to 1 year
  Mean values of the quantitative measures and proliferative ability will be calculated for each four time points and compared to determine the trajectory over time as described. In addition, the repeated measures for quantitative measures will be displayed graphically with individual trajectories. The linear mixed model will be performed to identify predictors (e.g., sex) that are associated with the quantitative measures. Furthermore, the generalized estimating equations model with the logit link and binomial distribution will be used to identify predictors for qualitative measures (e.g., prol
The quantity of cells determined by flow cytometry | Up to 1 year
  Mean values of the quantitative measures and proliferative ability will be calculated for each four time points and compared to determine the trajectory over time as described. In addition, the repeated measures for quantitative measures will be displayed graphically with individual trajectories. The linear mixed model will be performed to identify predictors (e.g., sex) that are associated with the quantitative measures. Furthermore, the generalized estimating equations model with the logit link and binomial distribution will be used to identify predictors for qualitative measures (e.g., prol

SECONDARY OUTCOMES:
Response of the tetanus toxoid vaccine-specific IgG antibody | At 28 days following tetanus toxoid vaccination
  Baseline and day 28 geometric mean titers (GMTs) will be calculated for hepatitis A or B and tetanus. GMTs for patients undergoing vaccination pre- and post-treatment will be performed. The difference in 28 day GMT between pretreatment and posttreatment will be compared using the paired t test. Analysis of covariance will be used to identify predictors that are associated with the change of 28 day difference in GMT. Seroconversion or a 4-fold rise in GMT from baseline to day 28 will be determined for pre and post treatment patient cohorts. Seroconversion proportion will be compared against kno
Vaccine-specific total antibody response after hepatitis A vaccination. In hepatitis A exposed patients, hepatitis B will be used. | At 28 days post hepatitis A vaccination
  Baseline and day 28 geometric mean titers (GMTs) will be calculated for each vaccine (i.e. hepatitis A or B and tetanus). GMTs for patients undergoing vaccination pre- and post-treatment will be performed. The difference in 28-day GMT between pre-treatment and post-treatment will be compared using the paired-t test. Analysis of covariance will be used to identify predictors that are associated with the change of 28-day difference in GMT. Seroconversion or a 4-fold rise in GMT from baseline to day-28 will be determined for pre- and post-treatment patient cohorts. Seroconversion proportion will

OTHER OUTCOMES:
Frequency of viral infection | Up to 1 year
  The distribution will be plotted using a histogram. Assessment of influenza vaccine immunogenicity will be performed. GMTs will be calculated at baseline and day 28. Seroconversion (i.e. 4-fold rise in GMT from baseline to day 28) will be determined. Proportions will be binned according to the timing of influenza vaccination: (1) pre-treatment, (2) during radiation, (3) during adjuvant chemotherapy, and (4) post-treatment. Seroconversion proportion within each time point will be compared against known normal using a one proportion test.
Overall survival (OS) | Date of surgery to death from any cause, assessed up to 14 months
  The Kaplan Meier method will be used to estimate OS probability and median time of survival along with 95% confidence interval. Proportional hazards models will be used to assess for associations between mortality and baseline quantitative immunologic values, baseline qualitative immunologic function, and baseline and post-treatment seroconversion to each vaccine (treated as a time dependent variable). All p-values will be reported as two-sided.
Titer of the influenza vaccine-specific IgG antibody | At 28 days following vaccination with the trivalent inactivated influenza vaccine
  Baseline and day 28 geometric mean titers (GMTs) will be calculated for hepatitis A or B and tetanus. GMTs for patients undergoing vaccination pre- and post-treatment will be performed. The difference in 28 day GMT between pretreatment and posttreatment will be compared using the paired t test. Analysis of covariance will be used to identify predictors that are associated with the change of 28 day difference in GMT. Seroconversion or a 4-fold rise in GMT from baseline to day 28 will be determined for pre and post treatment patient cohorts. Seroconversion proportion will be compared against kno

CONTACTS AND LOCATIONS:
Overall Officials: Roy Strowd, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Comprehensive Cancer Center of Wake Forest University, Winston-Salem, North Carolina, United States